CLINICAL TRIAL: NCT00439062
Title: Treatment of Rheumatoid Arthritis With Roxithromycin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nazilli State Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RA-89861966
Record Dates: First submitted 2007-02-20; First posted 2007-02-22 (Estimated); Last update posted 2007-02-22 (Estimated); Status verified 2007-02

CONDITIONS: Rheumatoid Arthritis
Keywords: Roxithromycin,Rheumatoid arthritis,Macrolides
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Roxithromycin

INTERVENTIONS:
Drug: Roxithromycin

SUMMARY:
The purpose of this study is to evaluate the clinical efficacy, safety, and tolerability of roxithromycin in patients with rheumatoid arthritis.

DETAILED DESCRIPTION:
This was 6-month, monocentre, randomized, double-blind, placebo-controlled study. We treated 100 patients with rheumatoid arthritis with either once-daily oral roxithromycin (300 mg) or daily oral placebo for 6 months. The primary efficacy variable was the percentage of patients who had a 20 percent improvement according to American College of Rheumatology (ACR) criteria (an ACR 20 response) at six months. Secondary outcome measures were 50 percent improvement and 70 percent improvement according to ACR criteria (an ACR 50 response and an ACR 70 response, respectively).

ELIGIBILITY:
Inclusion Criteria:RA according to the 1987 American Rheumatism Association criteria19, age between 18 and 70 years. Patients were required to have had an inadequate response to one to four DMARDs (such as azathioprine, methotrexate, sulfasalazine, penicillamine, hydroxychloroquine, or oral or injectable gold); an inadequate response was defined as discontinuation of therapy because of lack of effect. If patients were receiving DMARDs, they were required to complete a DMARD washout period that lasted at least 1 month before starting study drug treatment; no DMARDs were permitted during the study. Patients who were receiving nonsteroidal antiinflammatory drugs, prednisone (at 10 mg daily or less), or both were eligible if the doses had been stable for at least four weeks before the study period and continued to be stable during the study period. Patients were not allowed to receive intra-articular corticosteroids.

Patients had to have active disease at enrollment (before the DMARD washout period), defined as 12 or more tender joints, 10 or more swollen joints, and at least one of the following: erythrocyte sedimentation rate(ESR) of at least 28 mm/hr, C-reactive protein(CRP) level greater than 2.0 mg/dL, or morning stiffness for at least 45 minutes.

-

Exclusion Criteria:

* A negative pregnancy test result was required for non-menopausal female patients. In female patients of childbearing potential a urine pregnancy test was done at baseline and any pregnant women were excluded. Other exclusion criteria included impaired hepatic enzyme tests, impaired renal function, chronic/recurrent infection (e.g., chronic bronchitis, recurrent sinusitis), other infections(e.g., Borrelia burgdorferi, Chlamydia trachomatis, Ureaplasma) , history of adverse reactions to macrolides, roxithromycin, or similar antibiotics.

A patient could be withdrawn from the trial at any time after enrollment for the following reasons: the patient's request, severe or life-threatening adverse event, or inadequate control of arthritis symptoms (>50 percent increase in the total number of swollen or tender joints) necessitating an increase in the systemic corticosteroid dosage or reinstitution of therapy with disease-modifying antirheumatic drugs.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2006-06; Study Completion 2006-06

PRIMARY OUTCOMES:
The primary efficacy variable was the percentage of patients who had a 20 percent improvement according to American College of Rheumatology (ACR) criteria (an ACR 20 response) at six months.

SECONDARY OUTCOMES:
Secondary outcome measures were 50 percent improvement and 70 percent improvement according to ACR criteria (an ACR 50 response and an ACR 70 response, respectively).

CONTACTS AND LOCATIONS:
Overall Officials: Mesut Ogrendik, MD, Principal Investigator — Nazilli State Hospital
Locations (1):
- Nazilli State Hospital, Nazilli, Aydın, Turkey (Türkiye)

REFERENCES:
- [Derived] Ogrendik M, Karagoz N. Treatment of rheumatoid arthritis with roxithromycin: a randomized trial. Postgrad Med. 2011 Sep;123(5):220-7. doi: 10.3810/pgm.2011.09.2478. PMID 21904105